CLINICAL TRIAL: NCT01508455
Title: A Phase II/III, Open-Label, Multicenter, Safety, and Efficacy Study of Dexmedetomidine in Preterm Subjects Ages ≥28 Weeks to <36 Weeks Gestational Age
Brief Title: Open-Label, Safety, and Efficacy Study of Dexmedetomidine in Preterm Subjects Ages ≥28 Weeks to <36 Weeks Gestational Age
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEX-11-06
Record Dates: First submitted 2012-01-05; First posted 2012-01-12 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2015-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Fentanyl; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexmedetomidine (Experimental): Dexmedetomidine Load 0.2 mcg/kg over 10 or 20 min Dexmedetomidine Maintenance 0.2 mcg/kg/hr (at least 6 and up to 24 hours)
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam; Drug: Fentanyl; Drug: Morphine

INTERVENTIONS:
Drug: Dexmedetomidine
Drug: Midazolam
Drug: Fentanyl
Drug: Morphine

SUMMARY:
The primary objective of this study is to characterize the safety, and efficacy of Dexmedetomidine (DEX) administered as an intravenous (IV) loading dose followed by a continuous IV infusion in preterm subjects, ages ≥ 28 weeks through < 36 weeks gestational age.

ELIGIBILITY:
Inclusion Criteria:

1. Initially intubated and mechanically ventilated pediatric subjects in an intensive care setting anticipated to require at least 6 hours of continuous IV sedation.
2. Age: subjects must fit the following age range at screening:

   Preterm subjects ≥28 weeks through <36 weeks, gestational age;

   Note: Gestational age (in weeks) will be calculated as follows: the time elapsed between the first day of the last menstrual period and the day of enrollment.
3. Weight: subject's weight at the time of enrollment must be >1000 g.
4. Subject's parent(s) or legal guardian(s) has/have voluntarily signed and dated the informed consent document approved by the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).

Exclusion Criteria:

1. Neonate subjects with neurological conditions that prohibit an evaluation of sedation such as:

   * Diminished consciousness from increased intracranial pressure.
   * The presence of catastrophic brain injury or other severe mental disorders that would make responses to sedatives unpredictable and/or measurement of the N-PASS unreliable.
   * Subjects with immobility from neuromuscular disease or continuous infusion of neuromuscular blocking (NMB) agents.
2. Subjects with second degree or third degree heart block unless subject has a pacemaker or pacing wires are in situ.

   Note: If subject's status-post Cardio Pulmonary Bypass (CPB) was managed without pacing wires in situ, the subject must not be suspected to be in second degree or third degree heart block at the time of DEX administration.
3. HR < 120 bpm prior to the initiation of DEX.
4. Exposure to any investigational drug within 30 days prior to DEX administration.
5. Previous exposure to DEX as part of an investigational study.
6. In subjects that are ex-utero for less than 72 hours, a maternal history of poly-substance drug abuse, based upon the Investigator's clinical judgment.
7. At the discretion of the Investigator, subjects in whom the risk of DEX treatment is expected to exceed its benefits.
8. Subjects who have a known allergy or contraindication to fentanyl, morphine, MDZ, DEX, or other α-2 agonists.
9. Requirement for medications other than DEX, MDZ, morphine, or fentanyl for sedation and pain control.
10. Screening ALT levels >115 U/L.

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Louisville, Kentucky
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Morgantown, West Virginia

REFERENCES:
- [Derived] Chrysostomou C, Schulman SR, Herrera Castellanos M, Cofer BE, Mitra S, da Rocha MG, Wisemandle WA, Gramlich L. A phase II/III, multicenter, safety, efficacy, and pharmacokinetic study of dexmedetomidine in preterm and term neonates. J Pediatr. 2014 Feb;164(2):276-82.e1-3. doi: 10.1016/j.jpeds.2013.10.002. Epub 2013 Nov 14. PMID 24238862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Neonatal subjects enrolled from 3 centers in the United States
Period: Overall Study
Arm/Group | Dexmedetomidine
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects that received study drug.
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks]
  Age Continuous | 0.8 (1.36)
  Age Continuous: units: Gestational Age | 32.5 (2.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Requiring Rescue Midazolam for Sedation
Time Frame: During the study drug administration (ie., loading dose 10 or 20 minutes and maintenance infusion minimum of 6 hours up to 24 hours) and during the post drug administration (up to 24 hours).
Population: All Subjects who received study drug for at least 6 hours
Measure: Number; unit: percentage of participants
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 6
percentage of participants | 0

2. Secondary Outcome: Incidence of Rescue Medication (Fentanyl or Morphine) Use for Analgesia During DEX Infusion
Time Frame: as for outcome 1
Population: All subjects who received DEX for at least 6 hours formed the Efficacy Evaluable Population.
Measure: Number; unit: participant
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 6
participant | 1

3. Secondary Outcome: Amount of Rescue Medication (Midazolam) for Sedation During Dexmedetomidine Infusion
Time Frame: as for outcome 1
Population: No participants analyzed for this assessment since none required rescue Midazolam for sedation.
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 0

4. Secondary Outcome: Amount of Rescue Medication for Analgesia During DEX Infusion
Time Frame: as for outcome 1
Population: Number of subject who received rescue medication for analgesia during DEX infusion
Measure: Number; unit: mcg/kg
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 1
mcg/kg | 1

5. Secondary Outcome: Time Spent With a Total N-PASS Score >3 During DEX Infusion
Description: The N-PASS score >3 indicates adequately sedated and not manifesting signs of pain/agitation.
Time Frame: Predose, loading dose (LD) 5 & 10mins/if LD is 20mins (5, 10, 15 & 20mins); maintenance infusion: 0 min, every 15mins (1st hr); every 30mins (2hrs), then hourly; within 5mins of DEX discontinuation; 5mins pre and post rescue medication
Population: All subjects who received DEX for at least 6 hours formed the Efficacy Evaluable Population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 6
Hours | 0.44 (0.769)

6. Secondary Outcome: Time to Successful Extubation
Time Frame: From the start of study drug infusion to the study completion/withdrawal (Approximately 48 hours)
Population: Subjects who had successful extubation alone (n=5) were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 5
Hours | 37.3 [23.083 to 97.833]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events
Description: Treatment Emergent defined as start of study drug to 24 hours after discontinuation of study drug
Arm/Group | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=6)
Umbilcal hernia (Gastrointestinal disorders) | 1 (1)
Hypernatraenia (Metabolism and nutrition disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No